CLINICAL TRIAL: NCT07393958
Title: Experimental Study of Quality of Life in Patients With Endometriosis and Pelvic Pain Treated With Doliral Dietary Supplementation Versus Placebo.
Brief Title: Impact of Food Supplementation on Quality of Life in Patients With Endometriosis and Pelvic Pain.
Acronym: ENDOLIRAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arafarma Group, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ARA-EXP/DOL-2025-01
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Endometriosis (Diagnosis)
Keywords: pain; QoL; food supplement
MeSH Terms: conditions — Endometriosis; Disease; Pain | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Food supplement-Doliral) (Experimental): Patient takes one buccal tablet per day.
  Interventions: Dietary Supplement: Food supplement (T1675)
- Control (Placebo) (Placebo Comparator): Patient takes one buccal tablet per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement (T1675) — Doliral is the food supplement, which is the investigational product at this study.
  Arms: Experimental (Food supplement-Doliral)
Other: Placebo — Placebo is the control treatment.
  Arms: Control (Placebo)

SUMMARY:
This study examines whether the food supplement Doliral can improve quality of life and reduce pelvic pain in women with endometriosis, compared with placebo, over several weeks.

DETAILED DESCRIPTION:
Patients included into the study will be randomized into two treatment groups (30:30 patients). 30 patients will be treated with the food supplement and 30 patients will be treated with placebo. Both groups will be stratified by the presence or absence of hormonal therapy. Patients will be required to attend 6 study visits (selection visit, baseline or visit 0, and visits 1, 2, 3 and final or visit 4). Patients will complete a daily endometriosis symptom diary, which also includes a record of anti-inflammatory and paing medication use. Study treatment will be administred at Visit 0 or Baseline until Visit 4 or Final. At the study visits, patients will be requested to confirm the pain intensity through the VAS scale for different endometriosis pain types. They will be also requested to complete several questionnaires about quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age with diagnosed endometriosis stage I, II, or III, according to the American Society for Reproductive Medicine (ASRM) classification.
* Women with a diagnosis of endometriosis confirmed by laparoscopy or, in the absence of laparoscopy, by magnetic resonance imaging (MRI) and/or ultrasound.
* Presence of pelvic pain (VAS > 4) during the last three months.
* No indication for surgical intervention at the time of inclusion in the study.
* Patients who are able to provide informed consent.

Exclusion Criteria:

* Patients under 18 years of age.
* Use of analgesic or anti-inflammatory pharmacological treatment, except for ibuprofen at doses up to 600 mg/day or naproxen at doses up to 500 mg/day.
* Surgery within the year prior to inclusion, performed for therapeutic purposes related to the pathology under study.
* Initiation or discontinuation of hormone therapy within the three months prior to inclusion in the study.
* Patients with known allergy or hypersensitivity to Doliral®.
* Pregnant or breastfeeding patients.
* Patients on sick leave: > 1 year, or With no intention of returning to work, or Undergoing a disability or permanent incapacity assessment process.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
To measure the improvement of the quality of life. | From baseline visit to the final visit at 12 weeks.
  Patients complete EQ-5D-5L questionnaire at Day 1 (baseline visit), at 2 weeks (Visit 1), at 4 weeks (Visit 2), at 8 weeks (Visit 3) and at 12 weeks (Visit 4). This questionnaire measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression and health status. These five dimensions have 5 response levels: No problems, slight problems, moderate problems, severe problems and extreme problems. This questionnaire also has a Visual Analogue Scale from 0 (worse health status) to 100 (best health status).
To measure the improvement of the quality of life. | From baseline visit to the final visit at 12 weeks.
  Patients complete the Endometriosis Health Profile 30 Questionnaire at Day 1 (baseline visit), at 2 weeks (Visit 1), at 4 weeks (Visit 2), at 8 weeks (Visit 3) and at 12 weeks (Visit 4). This questionnaire evaluates six domains: pain, control and powerlessness, emotional well-being, social support and self-image. These scales are converted into a 0-100 score, 0 is best health status and 100 is worse quality of life.
To measure the improvement of the quality of life. | From baseline visit to the final visit at 12 weeks.
  Patients complete PGI-I (Patient Global Impression of Improvement) scale at Day 1 (baseline visit), at 2 weeks (Visit 1), at 4 weeks (Visit 2), at 8 weeks (Visit 3) and at 12 weeks (Visit 4). PGI-I is a Likert scale from 1 (significantly better) to 7 (significantly worse).
To measure the improvement in pain intensity. | From baseline visit to the final visit at 12 weeks.
  To describe the type and intensity of pain using a Visual Analogue Scale (VAS) at at Day 1 (baseline visit), at 2 weeks (Visit 1), at 4 weeks (Visit 2), at 8 weeks (Visit 3) and at 12 weeks (Visit 4). It is measured the change of these results from baseline visit to the final visit. Also patients complete a symptoms diary between visits. For each symptom, the patient will record intensity (on a scale from 1 to 10).

SECONDARY OUTCOMES:
Compare the reduction in the need for prescription and dosage of anti-inflammatory and analgesic pharmacological treatment. | From baseline visit to the final visit at 12 weeks.
  Patients will complete the use of inflammatory and analgesic pharmacological treatment (name, dose and time) in a diary between visits.
To measure the incidence of clinically relevant episodes | From Visit 1 (2 weeks) to Visit 4 or Final (12 weeks).
  To assess and destribe the type, intensity and relationship with investigational product of clinically relevant episodes at Day 1 (baseline visit), at 2 weeks (Visit 1), at 4 weeks (Visit 2), at 8 weeks (Visit 3) and at 12 weeks (Visit 4).

CONTACTS AND LOCATIONS:
Overall Officials: TAMARA RODRIGUEZ ARAYA, Dr, Principal Investigator — Hospital Clinic of Barcelona

IPD SHARING:
Plan to Share IPD: Undecided